CLINICAL TRIAL: NCT01704521
Title: Viral Kinetic Models of HCV Clearance in Hemophiliacs With Telaprevir
Brief Title: Viral Kinetics in HCV Clearance in Subjects With Hemophilia
Acronym: HCV/Hemophil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kenneth Sherman (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vertex Pharmaceuticals Incorporated (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kenneth Sherman, Kenneth E. Sherman, MD, PhD, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12053004; R34HL109334 (NIH)
Record Dates: First submitted 2012-10-05; First posted 2012-10-11 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Hepatitis C; Hemophilia
Keywords: Hepatitis C; HCV; Hemophilia
MeSH Terms: conditions — Hepatitis C, Chronic; Hemophilia A; Hepatitis C | interventions — Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lead-In (Active Comparator): Kinetic assessment of response guided treatment per standard of care with PegInterferon + Ribavirin for 4 weeks followed by 12 weeks of PegInterferon + Ribavirin + Telaprevir followed by variable duration of PegInterferon + Ribavirin
  Interventions: Drug: PegInterferon; Drug: Ribavirin; Drug: Telaprevir
- No Lead-in (Active Comparator): Kinetic assessment of response guided treatment per standard of care with PegInterferon + Ribavirin + Telaprevir for 12 weeks followed by variable duration of PegIntereron + Ribavirin
  Interventions: Drug: PegInterferon; Drug: Ribavirin; Drug: Telaprevir

INTERVENTIONS:
Drug: PegInterferon
Drug: Ribavirin
Drug: Telaprevir

SUMMARY:
This study will examine viral dynamic responses in subjects with chronic hepatitis C and hemophilia when treated with pegylated interferon + ribavirin and telaprevir.

DETAILED DESCRIPTION:
Previous clinical trials for treatment of chronic hepatitis C have excluded subjects with hemophilia from participating.

ELIGIBILITY:
Inclusion Criteria:

1. Hemophilia A or B
2. HCV RNA positive (PCR or branched-chain DNA Methods), Genotype 1 (a/b, mixed and unknown subtype)
3. Chronic HCV infection evidenced by HCV serology, HCV RNA or liver enzyme abnormalities present at least 6 months prior to enrollment
4. Liver biopsy or non-invasive marker that permits fibrosis staging within 12 months of enrollment. If a biopsy was not performed within 1 year, non-invasive markers may be utilized during screening period. Cirrhosis is not an exclusion factor
5. Age ≥ 18 years
6. Prior HCV treatment naïve or experienced
7. HCV viral load detectable during screening period
8. Absence of exclusion criteria
9. Sexually active subjects (both male and female) must agree and commit to the use of a medically acceptable form of contraception for the duration of the study and for 6 months following the last dose of study medication. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices or properly used barrier contraception.

Exclusion Criteria:

1. Hemoglobin <11
2. Pregnancy (during screening period or any time during treatment)

   1. females, that are planning to become pregnant or are breastfeeding
   2. males, whose partner is pregnant or is planning to become pregnant
3. HIV Infection
4. Prior History of:

   1. Hepatitis B (HBsAG negative - must have documentation of negative results within one year prior to enrollment or during screening period if not performed in that time window
   2. Homozygotic alpha-1-anti-trypsin (a1AT) deficiency - documentation of a1AT level <80 (at anytime prior to screening). If <80, phenotype testing should not demonstrate zz phenotype. All other phenotypes are not exclusionary,
   3. History of Homozygotic Genetic Hemochromatosis (at anytime prior to enrollment) with evidence of iron overload requiring phlebotomy,
   4. Autoimmune markers (antinuclear antibody (ANA) and/or antismooth muscle antibody (ASMA)) >1:160.
   5. Any other significant liver disease or process (to be determined by the investigator). Non-alcoholic fatty-liver disease (NAFLD) is not an exclusion.
5. History of Decompensated liver disease evidenced by any prior history of hepatic encephalopathy (Grade 2 or higher), ascites, variceal bleeding; Platelet count < 100,000
6. Active thyroid disease (OK if on thyroid replacement with normal thyroid-stimulating hormone (TSH); if TSH abnormal must have normal free thyroid index)
7. Chronic renal insufficiency, defined as creatinine clearance < 50 ml/min. (estimated by Modification of Diet in Renal Disease (MDRD) formula)
8. Life-threatening disease processes that could preclude completion of trial in opinion of investigator.
9. Any condition which the investigator feels will preclude safe completion of the treatment regimen including severe psychiatric disorders, active alcohol or recreational drug abuse.
10. Inability to provide informed consent.
11. Use of systemic corticosteroids or immunomodulatory drugs within 1 month (Nasal steroids are permitted.)
12. Uncontrolled seizure disorder (in opinion of investigator)
13. Concurrent autoimmune processes with active disease that may be exacerbated by interferon-based therapies (e.g. Crohn's Disease, Rheumatoid arthritis) in the opinion of the investigator. Psoriasis permitted if controlled with topical medications at the time of study enrollment.
14. Use of prohibited medications (as described in the telaprevir package insert) within 14 days of the first dose of study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Sherman, MD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- UC Physicians Company, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2013 through April 2014 at Digestive Diseases Research / University of Cincinnati
Groups:
- No Lead-in: No 4 week lead-in: Kinetic assessment of response guided treatment per standard of care with PegInterferon + Ribavirin + Telaprevir for 12 weeks followed by variable duration of PegInterferon + Ribavirin
Period: Overall Study
Arm/Group | Lead-In | No Lead-in
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-In | No Lead-in | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Median (Full Range); unit: years] | 53 [38 to 54] | 37 [27 to 47] | 47 [27 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virological Response at Week 12 (SVR12)
Description: Viral kinetic assessment using SVR 12 to either "lead-in" 4 weeks with PegInterferon + Ribavirin or no lead-in, followed by response guided therapy of 24 or 48 weeks based on viral response to treatment. Standard of care treatment stopping rules will be followed with assessment of viral response at week 12 of treatment.
Time Frame: Post-treatment at week 12
Population: See baseline characteristics
Measure: Number; unit: participants
Groups:
- No Lead-in: No 4 week lead-in: Kinetic assessment of response guided treatment per standard of care with PegInterferon + Ribavirin + Telaprevir for 12 weeks followed by variable duration PegInterferon + Ribavirin
Arm/Group | Lead-In | No Lead-in
Number analyzed (Participants) | 3 | 2
participants | 2 | 2

ADVERSE EVENTS:
Time Frame: Participants were assessed throughout their treatment intervention and through a 12 week followup period after completion of therapy, up to 60 weeks.
Description: Adverse events were only collected with regard to the affected organ system. Specific Adverse Event Terms are unknown.
Arm/Group | Lead-In | No Lead-in
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-In (N=3) | No Lead-in (N=2)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Not study drug related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-In (N=3) | No Lead-in (N=2)
General disorders (General disorders) | 3 (3) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) | 1 (1)
Skin and sucutaneous-tissue disorders (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 3 (3) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Cardiovascular disorders (Cardiac disorders) | 1 (1) | 0 (0)
Musculoskelatal disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Genitourinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Infections and infestations (Infections and infestations) | 2 (2) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No